CLINICAL TRIAL: NCT05937347
Title: Mindfulness and Cognitive Training Programs for Children with Attention Deficit Hyperactivity Disorder (ADHD): a Randomized, Controlled Trial (the NeuroMind Study)
Brief Title: Mindfulness and Cognitive Training Programs for Children with ADHD (the NeuroMind Study)
Acronym: NeuroMind
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Sant Joan de Déu (Other)
Collaborators: Universitat Autonoma de Barcelona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NeuroMind
Record Dates: First submitted 2023-05-29; First posted 2023-07-10 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2023-06

CONDITIONS: ADHD
Keywords: ADHD; Children; Mindfulness; Cognitive Training; Randomized Controlled Trial
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- TAU + UP4H (Experimental): UP4H is a face-to-face and virtual non-pharmacological program based on Mindfulness Training and Cognitive Training.
  Interventions: Behavioral: TAU + UP4H
- TAU + M4H (Active Comparator): M4H is a face-to-face non-pharmacological program based on Mindfulness Training.
  Interventions: Behavioral: TAU + M4H
- TAU + CT (Active Comparator): CT is a virtual non-pharmacological program based on Cognitive Training.
  Interventions: Behavioral: TAU + CT
- Treatment as Usual (TAU) (Active Comparator): Treatment as Usual (TAU) consisted of the prescribed drugs adapted to the ADHD symptomatic profile of each child.
  Interventions: Other: Treatment as Usual (TAU)

INTERVENTIONS:
Behavioral: TAU + UP4H — Group treatment protocol of 8 weeks (approximately 105 minutes per week, 75 of face-to-face and 30 of virtual intervention).
  Arms: TAU + UP4H
Behavioral: TAU + M4H — Group treatment protocol of 8 weekly 75 minute sessions (face-to-face intervention).
  Arms: TAU + M4H
Behavioral: TAU + CT — Group treatment protocol of 8 weekly 60 minutes sessions (virtual intervention).
  Arms: TAU + CT
Other: Treatment as Usual (TAU) — Standard pharmacological treatment usually provided to children with ADHD.
  Arms: Treatment as Usual (TAU)

SUMMARY:
The present project will evaluate through a Randomized Controlled Trial (RCT) with 5-month follow-up, the efficacy (5-month time horizon), adjunctive to TAU, of three 8-week interventions: a) the Mindfulness for Health program (i. e., M4H), b) a Cognitive Training (CT) program through NeuronUp platform and a program combining both (Mindfulness and Cognitive Training program, i. e., UP4H), a, as compared to TAU, in children (7-12 years old) with ADHD. In order to evaluate stability of clinical changes and to determine the mechanisms of action of the interventions studied, pre-post changes and at 5-months followup after the start of treatment will be evaluated in ADHD symptoms (inattention, hyperactivity, impulsivity), general functioning, clinical global impression, executive functions (verbal fluency, working memory, cognitive flexibility, inhibition), and comorbid symptoms (disruptive behavior, anxiety and depression) along with mindfulness skills. In the field of personalized treatment in ADHD, the design of the present study will also make it possible to establish whether certain baseline psychosocial and clinical characteristics may be associated with short- and medium-term clinical response to each of the treatments studied.

DETAILED DESCRIPTION:
Introduction: The NeuroMind study is aimed at assessing the efficacy of 3 interventions based on Mindfulness and/or Cognitive Training programs: a Mindfulness and Cognitive Training program (i. e., UP4H), a Mindfulness program (i. e., M4H) and a Cognitive Training program (i. e. CT). This study will evaluate the short- and mid-time efficacy of these 3 interventions for the first time in children with ADHD. The objectives of this 5-month RCT, are (i) to examine the efficacy of adding UP4H, M4H or CT to treatment-as-usual (TAU) for children (7-12 years old) with ADHD; (ii) to identify pre-post differences in ADHD symptoms (inattention, hyperactivity, impulsivity), in executive functions (verbal fluency, working memory, cognitive flexibility, inhibition), and in comorbid symptoms (disruptive behavior, anxiety and depression) in the four study arms and (iii) to analyze the role of the mindful attention awareness as a psychological process variable mediator of 5-month clinical outcomes. Methods and analysis: Participants will be 120 children with ADHD (7-12 years old) recruited at CSMIJ Sant Joan de Déu Terres de Lleida (Lleida, Spain), randomly allocated to one of the four study arms: TAU vs TAU+CT vs TAU+M4H vs TAU+UP4H. A comprehensive assessment to collect ADHD symptoms (inattention, hyperactivity, impulsivity), executive functions (verbal fluency, working memory, cognitive flexibility, inhibition), comorbid symptoms (disruptive behavior, anxiety and depression), mindful attention awareness, general functioning and clinical global impression will be conducted pre-intervention, post-intervention (8 weeks), and at 5-month follow-up. Linear mixed-effects model analyses, mediation analysis and sensitivity analyses will be conducted on the basis of intention-to-treat approach and according to whether the patients are completers, or whether they completed the majority of the sessions (75% attendance).

ELIGIBILITY:
Inclusion Criteria:

* Children of both sexes, between 7 and 12 years of age.
* Diagnosis of ADHD according to the DSM-5 criteria by a specialist and confirmed by the Kiddie-Schedule for Affective Disorders and Schizophrenia, Present and Lifetime Version (K-SADS-PL).
* ADHD medication dose is stable in the last 2 months or there is an informed decision on not taking ADHD medication.
* Children and parents have an adequate mastery of the Spanish language.
* Children and parents are available to meet all visits.
* Children's representatives (either parents or legal guardians) must understand the conditions of the study and sign the informed consent.
* Psychiatric comorbidities are allowed except psychosis, bipolar illness, active suicidality, untreated posttraumatic stress disorder or substance use (checked by the structured interview K-SADS-PL) , provided ADHD is the primary diagnosis in the child.
* Children have an IQ ≥ 80 checked by the Kaufman Brief Intelligence Test (K-BIT).

Exclusion Criteria:

* Diagnosis of Autism Spectrum Disorder (ASD) according to the DSM-5 criteria by a specialist or confirmed by the Social Communication Questionnaire (SCQ).
* Children who received psychological or psycho-educational treatment in the last 2 months or whose parents don't agree not to seek it during the study.
* Children have participated in a mindfulness programme in the past or the current year
* Children are participating in another clinical trial.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 122 (Actual)
Dates: Start 2023-07-20 (Actual); Primary Completion 2024-03-22 (Actual); Study Completion 2024-07-26 (Actual)

PRIMARY OUTCOMES:
ADHD symptoms (inattention, hyperactivity, impulsivity) | Change from baseline values at 5 months
  Conners' Parent Rating Scale-Revised (CPRS-R) Short form
ADHD symptoms (inattention, hyperactivity, impulsivity) | Change from baseline values at 5 months
  Conners Continuous Performance Test 3rd Edition (CPT-3)

SECONDARY OUTCOMES:
Executive functions (verbal fluency, working memory, cognitive flexibility, inhibition) | Change from baseline values at 5 months
  Neuropsychological Assessment of Executive Functions in Children (ENFEN)
Disruptive behavior, anxiety and depression | Change from baseline values at 5 months
  Child Behavior Checklist (CBCL)
Mindful attention awareness | Change from baseline values at 5 months
  Mindful Attention Awareness Scale Adapted for Children (MAAS-C). Total scores of the MAAS-C range from 15 to 90, where higher scores mean a better mindful attention awareness.
General functioning | Change from baseline values at 5 months
  Children's Global Assessment Scale (CGAS). Total scores of the CGAS range from 1 to 100, where higher scores means a better general functioning.
Clinical Global Impression | Change from baseline values at 5 months
  Clinical Global Impression Scale (CGI). Total scores of the CGI range from 0 to 7, where higher scores means a worse clinical global impression.
Anxiety | Change from baseline values at 5 months
  Screen for Child Anxiety Related Disorders (SCARED)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Huguet, PhD, Principal Investigator — CSMIJ Sant Joan de Déu Terres de Lleida; Albert Feliu, PhD, Principal Investigator — Universitat Autonoma de Barcelona
Locations (1):
- Fundació Privada per a la Recerca i la Docència Sant Joan de Déu (FSJD), Esplugues de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Badia-Aguaron T, Royuela-Colomer E, Pera-Guardiola V, Verges-Balasch P, Cebolla A, Luciano JV, Soler J, Feliu-Soler A, Huguet Miguel A. Combining mindfulness and cognitive training in children with attention deficit hyperactivity disorder: study protocol of a pilot randomized controlled trial (the NeuroMind study). Front Psychol. 2024 Feb 7;15:1291198. doi: 10.3389/fpsyg.2024.1291198. eCollection 2024. PMID 38384348